CLINICAL TRIAL: NCT05703308
Title: Outcome of Pregnancy in Poor Ovarian Responders by Intraovarian Administration of Autologous Menstrual Blood Derived-Mesenchymal Stromal Cells
Brief Title: Menstrual Blood Stem Cells in Poor Ovarian Responders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avicenna Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 99008-1023
Record Dates: First submitted 2023-01-15; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Poor Ovarian Response; Infertility, Female
Keywords: Poor Ovarian Responders; Menstrual Blood Stem cells; Infertility; Cell therapy; ICSI
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MenSCs group (Experimental): Study group, treated with autologous intra-ovarian MenSCs injection and monitored for spontaneous pregnancy for 3 months after intervention. ICSI was used in cases where the pregnancy did not occur naturally.
  Interventions: Biological: Autologous Menstrual Blood Stem Cells
- ICSI group (No Intervention): Control group, monitored for spontaneous pregnancy for 3 months after their last ovarian stimulation for ICSI or IVF. ICSI was used in cases where the pregnancy did not occur naturally.

INTERVENTIONS:
Biological: Autologous Menstrual Blood Stem Cells — The menstrual blood of patients in the MenSCs treatment group was collected in sterile menstrual cups on the second day of menstruation, and directly transferred to a class B clean room for MSC isolation and culture. All cell quality control studies were performed prior to the International Conference of Harmonization Q2 (ICH Q2) guidelines. The density of the final product was 20×106 cells/ml. 150 μl of the prepared suspension was injected intravaginally into each ovary of the patient under general anaesthesia
  Arms: MenSCs group

SUMMARY:
In this controlled trial, poor ovarian responder women will be treated with transplantation of autologous menstrual blood stem cells. The investigators will attempt to assess the safety and efficacy of this procedure for the treatment of infertility in POR patients compared to control group.

DETAILED DESCRIPTION:
With economic development, procreation delays have resulted in more women seeking medical help for infertility treatment. Because the quality and quantity of oocytes are affected by physiological age, despite advances in assisted reproductive technology (ART), managing infertility in women with poor ovarian response (POR) remains a daily challenge for physicians.

Adult mesenchymal stromal cell (MSC) therapy has gained particular interest in recent years because it may provide a supportive microenvironment for oocyte development from quiescent primordial follicles. Human MSC transplantation has been shown in preclinical studies to host ovaries and restore their function and structure premature ovarian failure (POF) animal models.

Because of their encouraging characteristics such as ease of access, high availability, monthly repeatability of sampling, less ethical considerations, lack of tumor-causing potential, protected property, and significant trans-differentiation capacity, endometrial-derived stromal cells have been considered in a wide range of studies since 2007. Menstrual blood-derived stromal cells (MenSCs), on the other hand, are derived from endometrial tissue and can be collected in a non-invasive manner, making them especially useful in the treatment of reproductive disorders. The investigators attempted to assess the safety and efficacy of intraovarian injection of MenSCs for the treatment of infertility in POR patients based on this evidence.

The results of this clinical trial's phases I and II indicated that Men-MSCs could be considered as a potential treatment to restore the fertility capability of POR women. Based on these findings, the investigators have designed a Phase III controlled trial of autologous MenSC therapy for patients with POR.

ELIGIBILITY:
Inclusion Criteria:

* Serum AMH < 0.1 ng/ml (at the screening visit and in the absence of OC or sex-steroid intake)
* Antral follicular count (AFC) in both ovaries < 4 (at screening visit and in the absence of OC or sex-steroid intake)
* Positive history of at least1 standard previous IVF-ET or ICSI-ET
* Normal thyroid hormones (TSH and FT4)
* Normal level of prolactin,
* Normal level of fasting blood sugar
* Normal Liver tests (SGOT, SGPT)
* Normal level of BUN, creatinine
* Negative Infectious tests (HIV, HCV, HBS Ag, VDRL)
* Normal coagulation factors (PT, PTT, BT, CT)
* Normal serum levels of sodium, potassium, calcium, phosphorus
* Negative history of endometrioma or other ovarian cysts
* Negative history of previous ovarian surgery
* Negative history of cancer
* Negative history of a known autoimmune disorder.

Exclusion Criteria:

* Positive history of hydrosalpinx or anatomical uterine disorders (In vaginal sonography or HSG)
* Severe male factors of their husbands (count <15 million/ml)

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2020-06-21 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2022-10-22 (Actual)

PRIMARY OUTCOMES:
Spontaneous pregnancy rate | 3 months after stem cell injection
  Number of participants that establish a spontaneous clinical pregnancy after stem cell injection
Pregnancy rate after ICSI | 4 weeks after embryo transfer
  Number of participants that establish a clinical pregnancy after embryo transfer

SECONDARY OUTCOMES:
Hormone levels | 2 and 4 months after stem cell injection
  Change from baseline in Anti-Müllerian hormone (AMH), serum follicle stimulating hormone (FSH), and antral follicle count (AFC)
Number of oocytes | Day 0 after follicle puncture
  Mean number of retrieved COCs per protocol
Number of MII oocytes | Day 0 after follicle puncture
  Mean number of metaphase II (MII) oocytes per protocol
Number of embryos | Day 3-5 after follicle puncture
  Mean number of embryos
Number of high quality embryos number | Day 3-5 after follicle puncture
  Grade A for cleavage stage embryo, >=3BB for blastocyst
Clinical pregnancy rate | 4 weeks after embryo transfer
  The incidence of gestational sac with heartbeat assessed by TVS
Biochemical pregnancy rate | 12-16 days after oocyte pick-up
  Incidence of serum beta-hCG test > 25 mIU/ml
Live birth rate | at a follow-up time of 30 days after delivery
  Incidence of the birth of at least one live newborn after 22 weeks of gestation
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | at a follow-up time after 1 year
  Incidence of adverse and serious adverse events with potential relationship to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Simin Zafardoust, MD, Study Director — Nanbiotechnology Research Center Avicenna Research Institute, ACECR, Tehran, Iran.; Somaieh Kazemnejad, Study Chair — Nanbiotechnology Research Center Avicenna Research Institute, ACECR, Tehran, Iran.; Mina Fathi Kazerooni, MD, PhD, Principal Investigator — Nanbiotechnology Research Center Avicenna Research Institute, ACECR, Tehran, Iran.
Locations (1):
- Avicenna Research Institute, Tehran, Iran

REFERENCES:
- [Derived] Zafardoust S, Kazemnejad S, Fathi-Kazerooni M, Darzi M, Sadeghi MR, Sadeghi Tabar A, Sehat Z. The effects of intraovarian injection of autologous menstrual blood-derived mesenchymal stromal cells on pregnancy outcomes in women with poor ovarian response. Stem Cell Res Ther. 2023 Nov 15;14(1):332. doi: 10.1186/s13287-023-03568-1. PMID 37968668